

| Title: UCC-23AC023 Statistical Analysis Plan Table shells | Page No. |
|-----------------------------------------------------------|-------------|
| Study Title: UCC-23AC023 PureWick Adolescent Study | Version No: |
| CIP/CPSP Version: 1.0 | 1.0 |

Template GFM-10082B

| PREPARED BY: | | |
|-----------------|---------------------|------------------|
| Susie Xiao | 30-Sept-2024 | SAP Version: 1.0 |
| (Printed Name): | Date: (DD-MMM-YYYY) | |



| Title: UCC-23AC023 Statistical Analysis Plan Table shells | Page No. |
|-----------------------------------------------------------|-------------|

# **Table of Contents**

| 1.0 | GENERAL GUIDANCE ON OUTPUT FORMAT | 4 |
|---|---|---|
| | 1.1 Document Headers and Footnotes | 4 |
| | 1.2 Presentation of Table Numbering and Titles Within Document | 4 |
| | 1.3 Output Format | 5 |
| 2.0 | SHELLS AND SPECIFICATIONS FOR TABLES | 6 |
| | 2.1 Demographic Data Summary Figures and Tables | 6 |
| | Table 1 Subject Disposition | 6 |
| | Table 2 Analysis Population | 6 |
| | Table 3 Demographics and Baseline Characteristics by Gender | 6 |
| | Table 4 Protocol Deviations | 8 |
| | 2.2 Efficacy Data Summary of Figures and Tables | 9 |
| | 2.2.1 Treatment summary | 9 |
| | Table 5 Treatment Summary by Void | 10 |
| | Table 6 Treatment Summary by Placement | 12 |
| | Table 7 Treatment Summary by Device | 14 |
| | 2.2.2 Primary Endpoint 1 - Capture Rate | 16 |
| | Table 8a Void Summary by Device | 16 |
| | Table 8b Capture Rate by Device | 16 |
| | Table 9a Void Summary by Device and Placement | 17 |
| | Table 9b Capture Rate by Device and Placement | 17 |
| | 2.2.3 Primary Endpoint 2 - Perception of Wetness | 18 |
| | Table 10 Perception of Wetness Summary by Device | 18 |
| | Table 11 Perception of Wetness Summary by Device and Placement | 18 |
| | 2.2.4 Secondary Endpoint 1 – Ease of Use Score | 19 |
| | Table 12 Participant Ease of Use Questionnaire, Common Questions for Both Devices | 19 |
| | Table 13 Participant Ease of Use Questionnaire, PureWick Flex Only Questions | 20 |
| | Table 14 HCP Ease of Use Questionnaire | 21 |
| | 2.2.5 Secondary Endpoint 2 – Overall Comfort Score | 22 |
| | Table 15 Participant Comfort Scale Survey | 22 |
| | 2.2.6 Secondary Endpoint 3 - IFU comprehension score | 23 |



Title: UCC-23AC023 Statistical Analysis Plan Table shells
Page No.

Study Title: UCC-23AC023 PureWick Adolescent Study
CIP/CPSP Version: 1.0

| Tem | plate GFM-10082B Table 16 Participant IFU Comprehension Survey | 23 |
|-----|----------------------------------------------------------------|----|
| | 2.3 Safety Data Summary of Figures and Tables | 24 |
| 3.0 | SHELLS AND SPECIFICATIONS FOR LISTINGS | 25 |
| | 3.1 Subject Data Listings | 25 |
| | 3.1.1 Screen Failure | 25 |
| | Listing 1 Screen Failures | 25 |
| | Listing 2 Randomization and Treatment Status | 25 |
| | Listing 3 End of Study Status | 25 |
| | Listing 4 Protocol Deviations | 26 |
| | 3.1.4 Patients excluded from the Efficacy Analysis | 26 |
| | Listing 5 Voids did not meet Evaluable Criteria | 26 |
| | 3.1.5 Demographics Data | 27 |
| | Listing 6 Demographic Data | 27 |
| | Listing 7 Treatment Details (Part 1) | 27 |
| | Listing 8 Treatment Details (Part 2) | 28 |
| | Listing 9 Treatment Details (Part 3) | 29 |
| | Listing 10 Capture Rate | 29 |
| | Listing 11 Participant - Perception of Wetness | 30 |
| | Listing 12 Participant Ease of Use – Both Device | 30 |
| | Listing 13 Participant Ease of Use – PureWick Flex Female only | 31 |
| | Listing 14 HCP Ease of Use | 31 |
| | Listing 15 Participant IFU | 32 |
| | Listing 16 Participant Comfort Scale Survey | 32 |
| | Listing 17 Adverse Events | 33 |
| | Listing 18 Serious Adverse Events | 33 |
| | 3.1.9 Device Deficiency | 34 |
| | Listing 19 Device Deficiencies | 34 |
| 4.0 | REFERENCES | 34 |
| 5.0 | VERSION HISTORY | 34 |



| Title: UCC-23AC023 Statistical Analysis Plan Table shells | Page No. |
|-----------------------------------------------------------|-------------|

#### 1.0 GENERAL GUIDANCE ON OUTPUT FORMAT

It is suggested that computer-generated output adhere to the following specifications.

#### 1.1 Document Headers and Footnotes

Unless otherwise specified, all computer-generated output should be produced in landscape mode. Required margins: at least 1.25 inches on top (the binding margin [or left for portrait output]), at least 1 inch on right, left, and bottom. All output should have the following header at top of page:

BD

CIP: UCC-23AC023

Population: Enrolled, PP, ITT, etc.

Page n of N

And the following as footnote:

Program name: xxxxx.sas

Data Source: ADSL, ADTL, ADDEV,

ADIMFD, etc.

Cutoff Date: DD-MMM-YYYY

Date DD-MMM-YYYY: hhmmss

#### 1.2 Presentation of Table Numbering and Titles Within Document

Each output should be identified by a numeral followed by the title. The study population should be identified on the line immediately following the title. (example below.)

Table No. Table Title

**Table Title continued (if necessary)** 

Study population

#### Other general table formatting:

- Column headings should in initial upper-case characters,
- For numeric variables, include "unit" in column heading when appropriate.
- Only these categories for which there are at least one (1) subject represented in one (1) or more groups should be included.
- Footnotes should be single spaced but separated by at least a double space from the bottom line of the table. The notes are aligned vertically by the left vertical border of the table.



| Title: UCC-23AC023 Statistical Analysis Plan Table shells | Page No. |
|-----------------------------------------------------------|-------------|

#### 1.3 Output Format

 The estimated mean, median and standard deviation (SD) for a set of values should be printed out to one more decimal place than the individual units of measurement.
 For example, for age, with raw data in whole years, the following precision would be used:

#### **Example Formatting Requirements**

| n | XX |
|-----------|-------------|
| Mean (SD) | xx.x (xx.x) |
| Median | XX.X |
| Min – Max | xx – xx |

- Percentage values should be printed with one digit to the right of the decimal point (e.g., 12.8%, 5.4%). Less-than signs "<0.1%" should be printed when values are >0.0% and <0.1% (not 0.0%).
- Missing data should be represented on subject listings as either a hyphen ("-") with a
  corresponding footnote ("- = unknown or not evaluated"), or as "N/A," or with footnote
  or description, whichever is appropriate.
- Dates should be printed in SAS DATE9. format ("DDMMMYYYY": 01JUL2000).
   Missing portions of dates should be represented on subject listings as dashes (--JUL2000). Dates that are missing because they are not applicable for the subject are output as "N/A", unless otherwise specified.
- Time should be printed in SAS TIME5.format ("HH:MM": 17:30). Missing portions of time should be represented on subject listings as dashes (--:30). Times that are missing because they are not applicable for the subject are output as "N/A", unless otherwise specified.
- Data in columns of a table should be formatted as follows:
  - Alphanumeric values are left-justified
  - o Whole numbers (e.g., counts) are right-justified
  - Numbers containing fractional portions are decimal aligned
- For tables displaying counts and percent:
  - A data column entry of "n (%)" in the template indicates that the "N" in each column header will be used as denominator, unless a note indicates a different denominator is to be used.
  - A data column entry of "n/N (%)" in the template indicates that the number of nonmissing data values will be used as the denominator, unless a note indicates a different denominator is to be used.



| Title: UCC-23AC023 Statistical Analysis Plan Table shells | Page No. |
|-----------------------------------------------------------|-------------|

#### 2.0 SHELLS AND SPECIFICATIONS FOR TABLES

2.1 Demographic Data Summary Figures and Tables

#### **Table 1 Subject Disposition**

Enrolled

| Number of Participants | |
|--------------------------|-----------------------|
| Enrolled | n |
| Eligibility met | n |
| Randomized | <b>N</b> <sub>1</sub> |
| Completed Study | n(%) |
| Discontinued prematurely | n(%) |
| Withdrawal of Consent | n(%) |
| Adverse Event | n(%) |
| Death | n(%) |
| Protocol Deviation | n(%) |
| Sponsor Decision | n(%) |
| Investigator decision | n(%) |
| Other | n(%) |

Programming note: Display reasons of discontinuation reported for at least one subject only. n(%) divided by  $N_1$ 

# **Table 2 Analysis Population**

Enrolled

| | Total |
|-----------------------|-------|
| Enrolled | n |
| Intent-to-Treat (ITT) | n |
| Per-Protocol (PP) | n |

# Table 3 Demographics and Baseline Characteristics by Gender

ITT

| | Female | Male | Overall |
|------------------------|-------------|-------------|-------------|
| | (N=xxx) | (N=xxx) | (N=xxx) |
| Age (Years) | | | |
| N | XXX | XXX | XXX |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X | XX.X |
| Min – Max | XX - XX | XX - XX | xx - xx |
| Ethnicity | | | |
| Hispanic or Latino | n (%) | n (%) | n (%) |
| Not Hispanic or Latino | n (%) | n (%) | n (%) |
| Not Reported | n (%) | n (%) | n (%) |
| Unknown | n (%) | n (%) | n (%) |
| Race | | | |

THIS SUBJECT MATTER IS RESTRICTED SOLELY FOR THE USE OF BECTON DICKINSON AND COMPANY AND ITS SUBSIDIARIES



| Title: UCC-23AC023 Statistical Analysis Plan Table shells | Page No. |
|-----------------------------------------------------------|-------------|

| 0082B | | | |
|--------------------------|---------------|---------------|---------------|
| White | n (%) | n (%) | n (%) |
| Black or African | n (%) | n (%) | n (%) |
| American | ` , | , , | , , |
| American Indian or | n (%) | n (%) | n (%) |
| Alaska Native | | | |
| Asian | n (%) | n (%) | n (%) |
| Native Hawaiian or Other | n (%) | n (%) | n (%) |
| Pacific Islander | | | |
| Not Reported | n (%) | n (%) | n (%) |
| Unknown | n (%) | n (%) | n (%) |
| Two or More Races | n (%) | n (%) | n (%) |
| Weight (Kg) | | | |
| N | XXX | XXX | XXX |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X | XX.X |
| Min – Max | XX - XX | XX - XX | XX - XX |
| Height (cm) | | | |
| N | XXX | xxx | XXX |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X | XX.X |
| Min – Max | XX - XX | XX - XX | XX - XX |
| BMI (kg/m <sup>2</sup> ) | | | |
| N | XXX | XXX | XXX |
| Mean (SD) | xx.xx (xx.xx) | xx.xx (xx.xx) | xx.xx (xx.xx) |
| Median | XX.XX | XX.XX | XX.XX |
| Min – Max | XX.X - XX.X | XX.X - XX.X | XX.X - XX.X |
| BMI <40 | n (%) | n (%) | n (%) |
| BMI >=40 | n (%) | n (%) | n (%) |



| Title: UCC-23AC023 Statistical Analysis Plan Table shells | Page No. |
|-----------------------------------------------------------|-------------|

#### **Table 4 Protocol Deviations**

ITT

| | Subject |
|---------------------------------------------------------|----------------|
| | (N=xxx) |
| Number of Subjects with at Least One Protocol Deviation | n(%) |
| Total Number of Protocol Deviations | N <sub>1</sub> |
| Deviation from Protocol Defined Procedure | n(%) |
| Clinical Assessment Not Done | n(%) |
| Randomization Error | n(%) |
| Informed Consent | n(%) |
| Safety Reporting | n(%) |
| Clinical Assessment Out of Window | n(%) |
| Other | n(%) |
| Total Number of Major Protocol Deviations | n(%) |
| Number of Subjects with at Least One Major Protocol | n(%) |
| Deviation | 11(70) |
| Deviation From Protocol Defined Procedure | n(%) |

Programming note: Percentage of deviations use  $N_1$  as denominator; Percentage of Subjects use N as denominator.



| Title: UCC-23AC023 Statistical Analysis Plan Table shells | Page No. |
|-----------------------------------------------------------|-------------|

Template GFM-10082B

#### 2.2 Efficacy Data Summary of Figures and Tables

#### 2.2.1 Treatment summary

Note that some questions on treatment CRF are device specific or placement specific: Self-placed void only:

Did the guardian/parent help the participant place the device? Was the device correctly connected to canister via collector tubing? Did HCP feel the catheter was correctly placed?

Was catheter repositioned by participant after placement?

PureWick Flex Female only:

Did the catheter move or become dislodged?

For percentages, the total number of non- missing data counts will be used as the denominator.



| Title: UCC-23AC023 Statistical Analysis Plan Table shells | Page No. |
|-----------------------------------------------------------|-------------|

Template GFM-10082B

# **Table 5 Treatment Summary by Void**

| | Void 1 | Void 2 |
|---|---|---|
| | (N = xx) | (N = xx) |
| Device Placed by | | |
| Self Placed | n/N(%) | n/N(%) |
| HCP | n/N(%) | n/N(%) |
| Did Subject Participate in Device Placement/Void Attempt | | |
| Yes | n/N(%) | n/N(%) |
| No | n/N(%) | n/N(%) |
| Any Signs of Injury or Irritation in The Perineal Region Prior to Device Placement | | |
| Yes | n/N(%) | n/N(%) |
| No | n/N(%) | n/N(%) |
| Was Device Placed | | |
| Yes | n/N(%) | n/N(%) |
| No | n/N(%) | n/N(%) |
| Device | | |
| PureWick Flex Female | n/N(%) | n/N(%) |
| PureWick Male | n/N(%) | n/N(%) |
| Did the Guardian/Parent Help the Participant Place the Device | | |
| Yes | n/N(%) | n/N(%) |
| No | n/N(%) | n/N(%) |
| Was the Device Correctly Connected to Canister via Collector Tubing | | |
| Yes | n/N(%) | n/N(%) |
| No | n/N(%) | n/N(%) |
| Did HCP feel the catheter was correctly placed | | |
| Yes | n/N(%) | n/N(%) |
| No | n/N(%) | n/N(%) |



Title: UCC-23AC023 Statistical Analysis Plan Table shells
Page No.

Study Title: UCC-23AC023 PureWick Adolescent Study
CIP/CPSP Version: 1.0

1.0

Template GFM-10082B

| Was Catheter Repositioned by Partic | apant After Placement | | |
|---|---|---|---|
| Yes | | n/N(%) | n/N(%) |
| No | | n/N(%) | n/N(%) |
| Did the Participant Have a Void | | | |
| Yes | | n/N(%) | n/N(%) |
| No | | n/N(%) | n/N(%) |
| Did the catheter move or become dis | slodged | | |
| Yes | | n/N(%) | n/N(%) |
| No | | n/N(%) | n/N(%) |
| Was There Any Leakage Observed b | by HCP After the Void | | |
| Yes | | n/N(%) | n/N(%) |
| No | | n/N(%) | n/N(%) |
| Are There Any Signs of Injury or Irrita | ation in the Perineal Region or Adverse Reactions After Device Removal | | |
| Yes | | n/N(%) | n/N(%) |
| No | | n/N(%) | n/N(%) |
| Pad Starting Weight (g) | | | |
| N | | xxx | xxx |
| Mean (SD) | | xx.x (xx.x) | xx.x (xx.x) |
| Median | | XX.X | XX.X |
| Min – Max | | xxx-xxx | xxx-xxx |
| Pad Final Weight (g) | | | |
| N | | xxx | xxx |
| Mean (SD) | | xx.x (xx.x) | xx.x (xx.x) |
| Median | | XX.X | XX.X |
| Min – Max | | xxx-xxx | xxx-xxx |
| Canister Starting Weight (g) | | | |
| N | | XXX | xxx |
| Mean (SD) | | xx.x (xx.x) | xx.x (xx.x) |
| Median | | XX.X | XX.X |
| Min – Max | | xxx-xxx | xxx-xxx |
| Caniser Final Weight (g) | | | |
| N | | xxx | xxx |
| Mean (SD) | | xx.x (xx.x) | xx.x (xx.x) |
| Median | Downloaded on 09 Sep 2025 | xx.x | XX.X |
| Min – Max | System Version Number 1.0 | xxx-xxx | xxx-xxx |



| Title: UCC-23AC023 Statistical Analysis Plan Table shells | Page No. |
|-----------------------------------------------------------|-------------|

Template GFM-10082B

# **Table 6 Treatment Summary by Placement**

| | Self Placed | HCP |
|---|---|---|
| | (N = xx) | (N = xx) |
| Void | | |
| 1 | n/N(%) | n/N(%) |
| 2 | n/N(%) | n/N(%) |
| Did Subject Participate in Device Placement/Void Attempt | | |
| Yes | n/N(%) | n/N(%) |
| No | n/N(%) | n/N(%) |
| Any Signs of Injury or Irritation in The Perineal Region Prior to Device Placement | | |
| Yes | n/N(%) | n/N(%) |
| No | n/N(%) | n/N(%) |
| Was Device Placed | | |
| Yes | n/N(%) | n/N(%) |
| No | n/N(%) | n/N(%) |
| Device | | |
| PureWick Flex Female | n/N(%) | n/N(%) |
| PureWick Male | n/N(%) | n/N(%) |
| Did the Guardian/Parent Help the Participant Place the Device | | |
| Yes | n/N(%) | N/A |
| No | n/N(%) | N/A |
| Was the Device Correctly Connected to Canister via Collector Tubing | | |
| Yes | n/N(%) | N/A |
| No | n/N(%) | N/A |
| Did HCP feel the catheter was correctly placed | | |
| Yes | n/N(%) | N/A |
| No | n/N(%) | N/A |



Title: UCC-23AC023 Statistical Analysis Plan Table shells Page No. 13 of 33 Study Title: UCC-23AC023 PureWick Adolescent Study Version No: 1.0

CIP/CPSP Version: 1.0

Template GFM-10082B

| Was Catheter Repositioned by Pa | articipant After Placement | | |
|---|---|---|---|
| Yes | and partition in additional | n/N(%) | N/A |
| No | | n/N(%) | N/A |
| Did the Participant Have a Void | | 1,1,1(11) | |
| Yes | | n/N(%) | n/N(%) |
| No | | n/N(%) | n/N(%) |
| Did the catheter move or become | dislodged | | |
| Yes | • | n/N(%) | n/N(%) |
| No | | n/N(%) | n/N(%) |
| Was There Any Leakage Observe | ed by HCP After the Void | · · · | , , |
| Yes | • | n/N(%) | n/N(%) |
| No | | n/N(%) | n/N(%) |
| Are There Any Signs of Injury or In | rritation in the Perineal Region or Adverse Reactions After Device | | |
| Yes | | n/N(%) | n/N(%) |
| No | | n/N(%) | n/N(%) |
| Pad Starting Weight (g) | | | |
| N | | XXX | XXX |
| Mean (SD) | | xx.x (xx.x) | xx.x (xx.x) |
| Median | | XX.X | XX.X |
| Min – Max | | XXX-XXX | XXX-XXX |
| Pad Final Weight (g) | | | |
| N | | XXX | XXX |
| Mean (SD) | | xx.x (xx.x) | xx.x (xx.x) |
| Median | | XX.X | XX.X |
| Min – Max | | XXX-XXX | XXX-XXX |
| Canister Starting Weight (g) | | | |
| N | | XXX | XXX |
| Mean (SD) | | xx.x (xx.x) | xx.x (xx.x) |
| Median | | XX.X | XX.X |
| Min – Max | | xxx-xxx | XXX-XXX |
| Caniser Final Weight (g) | | | |
| N | | XXX | XXX |
| Mean (SD) | Downloaded on 09 Sep 2025 | xx.x (xx.x) | xx.x (xx.x) |
| Median | System Version Number 1.0 | XX.X | XX.X |
| Min – Max | | XXX-XXX | XXX-XXX |



Page No.


Version No:

1.0

Template GFM-10082B

# **Table 7 Treatment Summary by Device**

| | PureWick Flex Female | PureWick Male |
|---|---|---|
| | (N = xx) | (N = xx) |
| Void | | |
| 1 | n/N(%) | n/N(%) |
| 2 | n/N(%) | n/N(%) |
| Device Placed by | | |
| Self Placed | n/N(%) | n/N(%) |
| HCP | n/N(%) | n/N(%) |
| Did Subject Participate in Device Placement/Void Attempt | | |
| Yes | n/N(%) | n/N(%) |
| No | n/N(%) | n/N(%) |
| Any Signs of Injury or Irritation in The Perineal Region Prior to Device Placement | | |
| Yes | n/N(%) | n/N(%) |
| No | n/N(%) | n/N(%) |
| Was Device Placed | | |
| Yes | n/N(%) | n/N(%) |
| No | n/N(%) | n/N(%) |
| Did the Guardian/Parent Help the Participant Place the Device | | |
| Yes | n/N(%) | n/N(%) |
| No | n/N(%) | n/N(%) |
| Was the Device Correctly Connected to Canister via Collector Tubing | | |
| Yes | n/N(%) | n/N(%) |
| No | n/N(%) | n/N(%) |
| Did HCP feel the catheter was correctly placed | | |
| Yes | n/N(%) | n/N(%) |
| No | n/N(%) | n/N(%) |



Title: UCC-23AC023 Statistical Analysis Plan Table shells
Page No.

Study Title: UCC-23AC023 PureWick Adolescent Study
CIP/CPSP Version: 1.0

1.0

Template GFM-10082B

| Was Catheter Repositioned by Participant After Placement | | |
|---|---|---|
| Yes | n/N(%) | n/N(%) |
| No | n/N(%) | n/N(%) |
| Did the Participant Have a Void | | |
| Yes | n/N(%) | n/N(%) |
| No | n/N(%) | n/N(%) |
| Did the catheter move or become dislodged | | |
| Yes | n/N(%) | N/A |
| No | n/N(%) | N/A |
| Was There Any Leakage Observed by HCP After the Void | | |
| Yes | n/N(%) | n/N(%) |
| No | n/N(%) | n/N(%) |
| Are There Any Signs of Injury or Irritation in the Perineal Region or Adverse Reactions After Device Removal | | |
| Yes | n/N(%) | n/N(%) |
| No | n/N(%) | n/N(%) |
| Pad Starting Weight (g) | | |
| N | xxx | XXX |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X |
| Min – Max | xxx-xxx | xxx-xxx |
| Pad Final Weight (g) | | |
| N | xxx | xxx |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X |
| Min – Max | xxx-xxx | xxx-xxx |
| Canister Starting Weight (g) | | |
| N | xxx | xxx |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X |
| Min – Max | xxx-xxx | xxx-xxx |
| Caniser Final Weight (g) | | |
| N . | xxx | xxx |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median Downloaded on 09 Sep 2025 | XX.X | XX.X |
| Min – Max System Version Number 1.0 | xxx-xxx | XXX-XXX |



| Title: UCC-23AC023 Statistical Analysis Plan Table shells | Page No. |
|-----------------------------------------------------------|-------------|

#### 2.2.2 Primary Endpoint 1 - Capture Rate

Weight of Captured Urine = Canister final weight — Canister starting weight

Weight of Urine Leak =  $Bed\ pad\ final\ weight - Bed\ pad\ starting\ weight$ 

Void Weight = Weight of Captured Urine + Weight of Urine Leak

Capture Rate =  $\frac{weight\ of\ captured\ urine \times 100\%}{weight\ of\ captured\ urine + weight\ of\ urine\ leak}$ 

Voids with weight (captured + leak) >= 10 g is considered evaluable.

Capture rate is calculated from evaluable voids only.

#### **Table 8a Void Summary by Device**

ITT

| | PureWick Flex | PureWick Male |
|---------------------|---------------|---------------|
| | Female | (N = xx) |
| | (N = xx) | , , |
| Captured Weight (g) | | |
| N | XXX | xxx |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X |
| Min – Max | XXX-XXX | xxx-xxx |
| Leaked Weight (g) | | |
| N | XXX | XXX |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | xx.x |
| Min – Max | XXX-XXX | xxx-xxx |
| Void Weight (g) | | |
| N | XXX | xxx |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X |
| Min – Max | XXX-XXX | XXX-XXX |
| Evaluable Void | n (%) | n (%) |

#### **Table 8b Capture Rate by Device**

ITT

| _ ITT | | |
|---|---|---|
| Capture Rate (Evaluable Voids Only) | PureWick Flex<br>Female Evaluable | PureWick Male<br>Evaluable |
| | $(N_1 = xx)$ | $(N_1 = xx)$ |
| Mean (SD) | xx.x% (xx.x%) | xx.x% (xx.x%) |
| Median | xx.x% | xx.x% |
| Min - Max | xx.x% | xx.x% |

THIS SUBJECT MATTER IS RESTRICTED SOLELY FOR THE USE OF BECTON DICKINSON AND COMPANY AND ITS SUBSIDIARIES



| Title: UCC-23AC023 Statistical Analysis Plan Table shells | Page No. |
|-----------------------------------------------------------|-------------|
| CID/CDSD Varaion: 1.0 | 1.0 |

Note: Voids with weight (captured + leak) >= 10 g is considered evaluable.

# **Table 9a Void Summary by Device and Placement**

IT٦

| | HCP | | | SelfPlaced | SelfPlaced | |
|---|---|---|---|---|---|---|
| Device | PureWick Flex Female (N = xx) | PureWick<br>Male<br>(N = xx) | HCP Overall (N = xx) | PureWick<br>Flex Female<br>(N = xx) | PureWick<br>Male<br>(N = xx) | SelfPlaced<br>Overall<br>(N = xx) |
| Captured Weight (g) | , | | | | | |
| N | xxx | xxx | XXX | xxx | xxx | XXX |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min – Max | xxx-xxx | xxx-xxx | XXX-XXX | xxx-xxx | xxx-xxx | xxx-xxx |
| Leaked Weight (g) | | | | | | |
| N | xxx | XXX | xxx | xxx | XXX | XXX |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min – Max | xxx-xxx | xxx-xxx | XXX-XXX | xxx-xxx | xxx-xxx | xxx-xxx |
| Void Weight (g) | | | | | | |
| N | xxx | xxx | XXX | xxx | xxx | XXX |
| Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min – Max | xxx-xxx | XXX-XXX | XXX-XXX | xxx-xxx | XXX-XXX | XXX-XXX |
| Evaluable Void | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |

#### **Table 9b Capture Rate by Device and Placement**

ITT

| 111 | | | | | | |
|---|---|---|---|---|---|---|
| | HCP | | | SelfPlaced | | |
| Capture Rate<br>(Evaluable Voids Only) | PureWick<br>Flex Female<br>Evaluable<br>(N <sub>1</sub> = xx) | PureWick<br>Male<br>Evaluable<br>(N <sub>1</sub> = xx) | HCP Overall<br>Evaluable<br>(N <sub>1</sub> = xx) | PureWick Flex Female Evaluable (N <sub>1</sub> = xx) | PureWick<br>Male<br>Evaluable<br>(N <sub>1</sub> = xx) | SelfPlaced Overall Evaluable (N <sub>1</sub> = xx) |
| Mean (SD) | xx.x%<br>(xx.x%) | xx.x%<br>(xx.x%) | xx.x%<br>(xx.x%) | xx.x%<br>(xx.x%) | xx.x%<br>(xx.x%) | xx.x%<br>(xx.x%) |
| Median | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% |
| Min - Max | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% | xx.x% |

Note: Voids with weight (captured + leak) >= 10 g is considered evaluable.



Title: UCC-23AC023 Statistical Analysis Plan Table shells
Page No.

Study Title: UCC-23AC023 PureWick Adolescent Study
CIP/CPSP Version: 1.0

1.0

Template GFM-10082B

2.2.3 Primary Endpoint 2 - Perception of Wetness

#### **Table 10 Perception of Wetness Summary by Device**

ITT

| | PureWick Flex<br>Female<br>(N = xx) | PureWick Male<br>(N = xx) |
|---|---|---|
| Void Type | | |
| After HCP Placement Void | n (%) | n (%) |
| After Self Placement Void | n (%) | n (%) |
| Questionnaire Completed | | |
| Yes | n (%) | n (%) |
| No | n (%) | n (%) |
| How Wet or Dry did You Feel after Your<br>Urination | | |
| 1- Extremely Wet | n/N(%) | n/N(%) |
| 2- Very Wet | n/N(%) | n/N(%) |
| 3- Somewhat Wet | n/N(%) | n/N(%) |
| 4- Slightly Wet but Acceptably Dry | n/N(%) | n/N(%) |
| 5- Dry | n/N(%) | n/N(%) |
| Mean(SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X |
| Min-Max | XX-XX | XX-XX |
| Did You Feel Leakage While Voiding<br>During Use of the Device | | |
| Yes | n/N(%) | n/N(%) |
| No | n/N(%) | n/N(%) |

# Table 11 Perception of Wetness Summary by Device and Placement

ITT

| | After HCP Placement Void | | | After Self Placement Void | | |
|---|---|---|---|---|---|---|
| | PureWick Flex<br>Female<br>(N = xx) | PureWick<br>Male<br>(N = xx) | After HCP<br>Overall<br>(N = xx) | PureWick<br>Flex<br>Female<br>(N = xx) | PureWick<br>Male<br>(N = xx) | After Self<br>Overall<br>(N = xx) |
| Questionnaire Completed | | | | | | |
| Yes | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| No | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| How Wet or Dry did You<br>Feel after Your Urination | | | | | | |
| 1- Extremely Wet | n/N(%) | n/N(%) | n/N(%) | n/N(%) | n/N(%) | n/N(%) |
| 2- Very Wet | n/N(%) | n/N(%) | n/N(%) | n/N(%) | n/N(%) | n/N(%) |
| 3- Somewhat Wet | n/N(%) | n/N(%) | n/N(%) | n/N(%) | n/N(%) | n/N(%) |
| 4- Slightly Wet but | n/N(%) | n/N(%) | n/N(%) | n/N(%) | n/N(%) | n/N(%) |

THIS SUBJECT MATTER IS RESTRICTED SOLELY FOR THE USE OF BECTON DICKINSON AND COMPANY AND ITS SUBSIDIARIES



Title: UCC-23AC023 Statistical Analysis Plan Table shells
Page No.

Study Title: UCC-23AC023 PureWick Adolescent Study

Page No.

CIP/CPSP Version: 1.0

1.0

Template GFM-10082B

| Acceptably Dry | | | | | | |
|---|---|---|---|---|---|---|
| 5- Dry | n/N(%) | n/N(%) | n/N(%) | n/N(%) | n/N(%) | n/N(%) |
| Mean(SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) | xx.x<br>(xx.x) | xx.x<br>(xx.x) | xx.x<br>(xx.x) |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Min-Max | xx-xx | xx-xx | XX-XX | xx-xx | xx-xx | xx-xx |
| Did You Feel Leakage While Voiding During Use of the Device | | | | | | |
| Yes | n/N(%) | n/N(%) | n/N(%) | n/N(%) | n/N(%) | n/N(%) |
| No | n/N(%) | n/N(%) | n/N(%) | n/N(%) | n/N(%) | n/N(%) |

#### 2.2.4 Secondary Endpoint 1 - Ease of Use Score

# Table 12 Participant Ease of Use Questionnaire, Common Questions for Both Devices

| ITT | | |
|---|---|---|
| | PureWick Flex Female | PureWick Male |
| | (N = xx) | (N = xx) |
| Questionnaire Completed | | |
| Yes | n (%) | n (%) |
| No | n (%) | n (%) |
| How Easy was the Placement of the Device? | | |
| 1-Very Difficult | n/N(%) | n/N(%) |
| 2-Somewhat Difficult | n/N(%) | n/N(%) |
| 3-Average Difficulty | n/N(%) | n/N(%) |
| 4-Somewhat Easy | n/N(%) | n/N(%) |
| 5-Very Easy | n/N(%) | n/N(%) |
| Mean(SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X |
| Min-Max | xx-xx | xx-xx |
| How Easy was the Removal of the Device? | | |
| 1-Very Difficult | n/N(%) | n/N(%) |
| 2-Somewhat Difficult | n/N(%) | n/N(%) |
| 3-Average Difficulty | n/N(%) | n/N(%) |
| 4-Somewhat Easy | n/N(%) | n/N(%) |
| 5-Very Easy | n/N(%) | n/N(%) |
| Mean(SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X |
| Min-Max | XX-XX | XX-XX |



| Title: UCC-23AC023 Statistical Analysis Plan Table shells | Page No. |
|-----------------------------------------------------------|-------------|
| CID/CDSD Vorsion: 1.0 | 1.0 |

# Table 13 Participant Ease of Use Questionnaire, PureWick Flex Only Questions

| TT Female | - |
|-------------------------------------------|-------------------------------|
| | PureWick Flex Female (N = xx) |
| I was Able to Connect the Device | |
| PureWick Flex FEC Tubing | |
| 1-Strongly Disagree | n/N(%) |
| 2-Disagree | n/N(%) |
| 3-Neutral | n/N(%) |
| 4-Agree | n/N(%) |
| 5- Strongly Agree | n/N(%) |
| Mean(SD) | xx.x (xx.x) |
| Median | XX.X |
| Min-Max | XX-XX |
| I was Able to Locate the Vent Hole on the | |
| PureWick Flex FEC | |
| 1-Strongly Disagree | n/N(%) |
| 2-Disagree | n/N(%) |
| 3-Neutral | n/N(%) |
| 4-Agree | n/N(%) |
| 5- Strongly Agree | n/N(%) |
| Mean(SD) | xx.x (xx.x) |
| Median | XX.X |
| Min-Max | XX-XX |
| I would be able to tell if the PureWick | |
| Flex FEC came out of place | |
| 1-Strongly Disagree | n/N(%) |
| 2-Disagree | n/N(%) |
| 3-Neutral | n/N(%) |
| 4-Agree | n/N(%) |
| 5- Strongly Agree | n/N(%) |
| Mean(SD) | xx.x (xx.x) |
| Median | XX.X |
| Min-Max | XX-XX |
| I would be able to tell if the PureWick | |
| Flex FEC was in the Correct Orientation | |
| 1-Strongly Disagree | n/N(%) |
| 2-Disagree | n/N(%) |
| 3-Neutral | n/N(%) |
| 4-Agree | n/N(%) |

THIS SUBJECT MATTER IS RESTRICTED SOLELY FOR THE USE OF BECTON DICKINSON AND COMPANY AND ITS SUBSIDIARIES



| Title: UCC-23AC023 Statistical Analysis Plan Table shells | Page No. |
|-----------------------------------------------------------|-------------|

xx.x (xx.x)

XX.X

XX-XX

Template GFM-10082B 5- Strongly Agree n/N(%) Mean(SD) xx.x (xx.x) Median XX.XMin-Max XX-XX I Would be Able to Curve the PureWick Flex FEC to Fit My Body 1-Strongly Disagree n/N(%) 2-Disagree n/N(%) 3-Neutral n/N(%) 4-Agree n/N(%) 5- Strongly Agree n/N(%)

# Table 14 HCP Ease of Use Questionnaire

Mean(SD)

Median

Min-Max

| HCP | 1 | 1 |
|---|---|---|
| | PureWick Flex Female PureWick | |
| | $(HCP N = xx) \qquad (HCP N =$ | |
| Questionnaire Completed | | |
| Yes | n (%) | n (%) |
| No | n (%) | n (%) |
| How Easy was the Placement of the Device? | | |
| 1-Very Difficult | n/N(%) | n/N(%) |
| 2-Somewhat Difficult | n/N(%) | n/N(%) |
| 3-Average Difficulty | n/N(%) | n/N(%) |
| 4-Somewhat Easy | n/N(%) | n/N(%) |
| 5-Very Easy | n/N(%) | n/N(%) |
| Mean(SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X |
| Min-Max | xx-xx | XX-XX |
| How Easy was the Removal of the Device? | | |
| 1-Very Difficult | n/N(%) | n/N(%) |
| 2-Somewhat Difficult | n/N(%) | n/N(%) |
| 3-Average Difficulty | n/N(%) | n/N(%) |
| 4-Somewhat Easy | n/N(%) | n/N(%) |
| 5-Very Easy | n/N(%) | n/N(%) |
| Mean(SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X |
| Min-Max | xx-xx | XX-XX |



| Title: UCC-23AC023 Statistical Analysis Plan Table shells | Page No. |
|-----------------------------------------------------------|-------------|

# 2.2.5 Secondary Endpoint 2 – Overall Comfort Score

# **Table 15 Participant Comfort Scale Survey**

ITT

| | PureWick Flex | PureWick |
|---|---|---|
| | Female | Male |
| | (N = xx) | (N = xx) |
| Questionnaire Completed | | |
| Yes | n (%) | n (%) |
| No | n (%) | n (%) |
| How Comfortable was the Placement? | , | , , |
| 1-Very Uncomfortable | n/N(%) | n/N(%) |
| 2-Uncomfortable | n/N(%) | n/N(%) |
| 3-Neither Comfortable Nor Uncomfortable | n/N(%) | n/N(%) |
| 4-Comfortable | n/N(%) | n/N(%) |
| 5-Very Comfortable | n/N(%) | n/N(%) |
| Mean(SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X |
| Min-Max | XX-XX | XX-XX |
| How Comfortable was the Device While Voiding? | | |
| 1-Very uncomfortable | n/N(%) | n/N(%) |
| 2-Uncomfortable | n/N(%) | n/N(%) |
| 3-Neither Comfortable Nor Uncomfortable | n/N(%) | n/N(%) |
| 4-Comfortable | n/N(%) | n/N(%) |
| 5-Very Comfortable | n/N(%) | n/N(%) |
| Mean(SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X |
| Min-Max | XX-XX | XX-XX |
| How Comfortable was the Removal of the External Catheter? | | |
| 1-Very uncomfortable | n/N(%) | n/N(%) |
| 2-Uncomfortable | n/N(%) | n/N(%) |
| 3-Neither Comfortable Nor Uncomfortable | n/N(%) | n/N(%) |
| 4-Comfortable | n/N(%) | n/N(%) |
| 5-Very Comfortable | n/N(%) | n/N(%) |
| Mean(SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X |
| Min-Max | XX-XX | XX-XX |
| How Likely Would You Recommend the External Catheter to Someone Else? | | |
| 1-Very Unlikely | n/N(%) | n/N(%) |
| 2-Unlikely | n/N(%) | n/N(%) |
| 3-Neither likely Nor Unlikely | n/N(%) | n/N(%) |
| 4-Likely | n/N(%) | n/N(%) |
| 5-Very Likely | n/N(%) | n/N(%) |

THIS SUBJECT MATTER IS RESTRICTED SOLELY FOR THE USE OF BECTON DICKINSON AND COMPANY AND ITS SUBSIDIARIES



| Title: UCC-23AC023 Statistical Analysis Plan Table shells | Page No. |
|-----------------------------------------------------------|-------------|

| Mean(SD) | xx.x (xx.x) | xx.x (xx.x) |
|----------|-------------|-------------|
| Median | XX.X | XX.X |
| Min-Max | xx-xx | XX-XX |

#### 2.2.6 Secondary Endpoint 3 - IFU comprehension score

# Table 16 Participant IFU Comprehension Survey

| | PureWick Flex | PureWick |
|-------------------------------------------|---------------|-------------|
| | Female | Male |
| | (N = xx) | (N = xx) |
| Questionnaire Completed | | |
| Yes | n (%) | n (%) |
| No | n (%) | n (%) |
| I Was Able to Understand and Follow the | | |
| Written Instructions | | |
| 1-Strongly Disagree | n/N(%) | n/N(%) |
| 2-Disagree | n/N(%) | n/N(%) |
| 3-Neutral | n/N(%) | n/N(%) |
| 4-Agree | n/N(%) | n/N(%) |
| 5- Strongly Agree | n/N(%) | n/N(%) |
| Mean(SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X XX.X | |
| Min-Max | xx-xx | xx-xx |
| I Was Able to Understand the Pictures in | | |
| the Instructions | | |
| 1-Strongly Disagree | n/N(%) | n/N(%) |
| 2-Disagree | n/N(%) | n/N(%) |
| 3-Neutral | n/N(%) | n/N(%) |
| 4-Agree | n/N(%) | n/N(%) |
| 5- Strongly Agree | n/N(%) | n/N(%) |
| Mean(SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X |
| Min-Max | XX-XX | XX-XX |
| I Was Able to Place the PureWick External | | |
| Catheter on Myself | | |
| 1-Strongly Disagree | n/N(%) | n/N(%) |
| 2-Disagree | n/N(%) | n/N(%) |
| 3-Neutral | n/N(%) | n/N(%) |
| 4-Agree | n/N(%) | n/N(%) |
| 5- Strongly Agree | n/N(%) | n/N(%) |
| Mean(SD) | xx.x (xx.x) | xx.x (xx.x) |
| Median | XX.X | XX.X |
| Min-Max | XX-XX | XX-XX |



Template GFM-10082B

2.3 Safety Data Summary of Figures and Tables

Adverse events will be listed.



| Title: UCC-23AC023 Statistical Analysis Plan Table shells | Page No. |
|-----------------------------------------------------------|-------------|

Template GFM-10082B

#### 3.0 SHELLS AND SPECIFICATIONS FOR LISTINGS

- 3.1 Subject Data Listings
- 3.1.1 Screen Failure

# **Listing 1 Screen Failures**

| n | ro | ı | 0 |
|---|----|---|----|
| Ш | ıU | П | ピし |

| Subject ID | Eligibility criteria not met |
|------------|------------------------------|

#### 3.1.2 Enrollment details

# **Listing 2 Randomization and Treatment Status**

Enrolled

| Subject ID | Eligibility Met | Randomized? | Date of Randomization | Randomization No. | Randomized Sequence |
|---|---|---|---|---|---|
| | | Yes | | | |
| | | No | | | |

# **Listing 3 End of Study Status**

| | | | | Date of death | Primary cause of |
|---|---|---|---|---|---|
| Subject ID | Date of Study Completion/Discontinuation | Status | Other, Specify | | death |



| Title: UCC-23AC023 Statistical Analysis Plan Table shells | Page No. |
|-----------------------------------------------------------|-------------|
| 3.1.3 Protocol Deviations | 26 of 33 |

Template GFM-10082B

# **Listing 4 Protocol Deviations**

ITT

| Subject<br>ID | Date of<br>Deviation | Nature of Deviation | Major Protocol<br>Deviation |
|---|---|---|---|

# 3.1.4 Patients excluded from the Efficacy Analysis

# Listing 5 Voids did not meet Evaluable Criteria

| | | Device Placed | | Did the Participant Have a<br>Void | Pad Starting | <br>Canister<br>Starting Weight | Canister Final<br>Weight (g) |
|---|---|---|---|---|---|---|---|
| Subject ID | Void | Ву | Device | | Weight (g) | (g) | |



| Title: UCC-23AC023 Statistical Analysis Plan Table shells | Page No. |
|-----------------------------------------------------------|-------------|

Template GFM-10082B

# 3.1.5 Demographics Data

# **Listing 6 Demographic Data**

ITT

| Subject ID | Informed<br>Consent Date | Age | Sex | Race | Ethnicity | Height<br>(cm) | U | BMI<br>(kg/m²) |
|---|---|---|---|---|---|---|---|---|
| | 10MAR2024 | | | | Not Hispanic Or Latino | 170.0 | 109.0 | 37.7 |

# 3.1.6 Individual Efficacy Response data

# **Listing 7 Treatment Details (Part 1)**

| Subject<br>ID | Void | Was<br>Device<br>Placed | Device<br>Placed by | Device | Did<br>Participant<br>Have a Void | Signs of<br>Irritation Prior<br>(If yes, specify) | Signs of<br>Irritation<br>After<br>(If yes,<br>specify) | Did the Catheter<br>Move/Dislodged | Any<br>Leakage<br>Observed<br>by HCP |
|---|---|---|---|---|---|---|---|---|---|
| | Void<br>1 | Yes | HCP | | | | | | |
| | Void<br>2 | Yes | SelfPlaced | | | | | | |
| | | | | | _ | | | _ | |



| Title: UCC-23AC023 Statistical Analysis Plan Table shells | Page No. |
|-----------------------------------------------------------|-------------|

Template GFM-10082B

# Listing 8 Treatment Details (Part 2)

| Subject<br>ID | Void | Was<br>Device<br>Placed | Device<br>Placed by | Device | Did Subject Participate in Device Placement/Void Attempt | Did the<br>Guardian/Parent<br>Help the<br>Participant<br>Place the Device | Was the Device Correctly Connected to Canister via Collector Tubing (If No, Reason; If Other, Specify) | Did HCP<br>Feel the<br>Catheter<br>was<br>Correctly<br>Placed | Was Catheter Repositioned by Participant After Placement |
|---|---|---|---|---|---|---|---|---|---|
| | Void 1 | Yes | HCP | | | | • | | |
| | Void 2 | Yes | SelfPlaced | | | | | | |



Template GFM-10082B

# **Listing 9 Treatment Details (Part 3)**

ITT

| Subject<br>ID | Void | Was<br>Device<br>Placed | Device<br>Placed by | Device | Pad Starting Weight (g) | Pad Final<br>Weight (g) | Canister<br>Starting Weight<br>(g) | Canister Final<br>Weight (g) |
|---|---|---|---|---|---|---|---|---|
| | Void 1 | | | | | | | |
| | Void 2 | | | | | | | |

# **Listing 10 Capture Rate**

| Subject<br>ID | Void | Device<br>Placed by | Device | Leaked Weight | Captured<br>Weight (g) | Void Weight (g) | Evaluable | Capture Rate (%) |
|---|---|---|---|---|---|---|---|---|
| | Void 1 | | | | | | Yes | |
| | Void 2 | | | | | | No | N/A, Not<br>Evaluable |



Template GFM-10082B

# **Listing 11 Participant - Perception of Wetness**

ITT

| Subject<br>ID | Void | Device | Void Type | Questionnaire<br>Completed | How<br>Wet or Dry did<br>You Feel After<br>Your Urination | Comments if selected 1/2/3 | Did you Feel<br>Leakage While<br>Voiding |
|---|---|---|---|---|---|---|---|
| | Void 1 | | | | 1-Extremely Wet | | Yes |
| | Void 2 | | | | | | |

1.0

#### **Listing 12 Participant Ease of Use – Both Device**

| Subject ID | Questionnaire<br>Completed | Device | How Easy was the Placement of the Device | How Easy was the<br>Removal of the Device |
|---|---|---|---|---|
| • | | PureWick<br>Flex Female | 1-Very Difficult | |
| | | PureWick<br>Male | | |



Template GFM-10082B

# Listing 13 Participant Ease of Use – PureWick Flex Female only

ITT

| Subject<br>ID | Able to Connect<br>the Device<br>Tubing (If 1/2/3,<br>comments) | Able to Locate<br>the Vent Hole (If<br>1/2/3,<br>comments) | Able to Tell if<br>Came Out of Place<br>(If 1/2/3,<br>comments) | Able to Tell if in Correct<br>Orientation (If 1/2/3,<br>comments) | Able to Curve to Fit (If 1/2/3, comments) |
|---|---|---|---|---|---|
| | 1- Strongly | | | | |
| | Disagree<br>(xxxxx) | | | | |
| | (^^^ | | | | |

# **Listing 14 HCP Ease of Use**

| | _ | | • | |
|---|---|---|---|---|
| HCP Initials | Questionnaire<br>Completed | Device | How Easy was the<br>Placement of the Device | How Easy was the Removal of the Device |
| | | PureWick Flex Female | 1-Very Difficult | 5-Very Easy |
| | | PureWick Male | | |



| Title: UCC-23AC023 Statistical Analysis Plan Table shells | Page No. |
|-----------------------------------------------------------|-------------|

Template GFM-10082B

# **Listing 15 Participant IFU**

ITT

| Subject ID | Questionnaire<br>Completed | Device | Able to Understand Written Instructions (If 1/2/3, comments) | Able to Understand<br>Pictures Instructions<br>(If 1/2/3, comments) | Able to Place on<br>Myself (If 1/2/3,<br>comments) |
|---|---|---|---|---|---|
| _ | | PureWick | | | |
| | | Flex | | | |
| | | Female | 1-Strongly Disagree (xxxxxx) | | |
| | | PureWick | | | |
| | | Male | | | |

# Listing 16 Participant Comfort Scale Survey

| Subject<br>ID | Questionnaire<br>Completed | Device | How Comfortable was the Placement | How Comfortable was the device while voiding | How Comfortable was the Removal | How Likely to<br>Recommend |
|---|---|---|---|---|---|---|
| | | | | 1-Very | | |
| | | | 2-Uncomfortable | Uncomfortable | 5-Very Comfortable | 4-Likely |



Template GFM-10082B

#### **Listing 17 Adverse Events**

ITT

| Subject<br>ID | AE(Reported)/SOC/PT | Start Date<br>/ End Date | Outcome of AE | Severity | Relation to<br>Study<br>Device | Relation to | SAE | | Additional<br>Details |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | Yes/xxx | Yes/xxx | | Yes/No | |
| | | | | | No | | | | |

Page No. **33 of 33** 

Version No:

# **Listing 18 Serious Adverse Events**

| | | | Result | Life | If Require o<br>Hospitalizat | | Permanent<br>Impairment<br>of a Body<br>Structure<br>or Function | Necessitates<br>Medical or<br>Surgical<br>Intervention | Fetal Distress, Fetal Death, Congenital Anomaly or Birth Defect | Meet Definition of Serious Health Threat |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | AE(Reported)/SOC/PT | Start<br>Date | in<br>Death | Threatening<br>or Injury | Admission<br>Date | Discharge<br>Date | | | | |



Template GFM-10082B

# 3.1.9 Device Deficiency

# **Listing 19 Device Deficiencies**

ITT

| | Date of | | | | | | | | AE | | Meet Definition of |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Device | Time of | Device | | | | | Device | Associated | Could the Device | Serious Health |
| Subject | Deficien | Device | Name/identi | Failure | | Additiona | Lot | Used to | with Device | Deficiency Meet | Threat |
| ID <sup>°</sup> | cies | Deficiencies | fier | Code | Details | l Details | Number | Treat Subject | Deficiencies | SADE | |
| | DDMMY | | | | | | | Yes/No | Yes/No | | |
| | YY | | | | | | | | | | |

#### 4.0 REFERENCES

N/A

# 5.0 VERSION HISTORY

| Vers. # | Date | Change Owner | Description of Change(s) |
|---------|-----------|--------------|--------------------------|
| 1.0 | 9/30/2024 | | Original |



# Signature Page for VV-TMF-319540 v1.0

| Reason for signing: Finalize | Name: Ajesh Raju<br>Role: Clinical Project Management<br>Date of signature: 30-Sep-2024 20:06:09 GMT+0000 |
|---|---|
| Reason for signing: Finalize | Name: Swathi Vasireddi<br>Role: Clinical Statistical Programmer<br>Date of signature: 30-Sep-2024 20:44:55 GMT+0000 |
| Reason for signing: Finalize | Name: Yanchang Zhang<br>Role: Clinical Statistician<br>Date of signature: 01-Oct-2024 16:10:09 GMT+0000 |
| Reason for signing: Finalize | Name: Danielle Redmond<br>Role: Medical Affairs Core Team Member<br>Date of signature: 02-Oct-2024 14:19:49 GMT+0000 |
| Reason for signing: Finalize | Name: Shujie (Susie) Xiao<br>Role: Clinical Statistician<br>Date of signature: 02-Oct-2024 20:43:35 GMT+0000 |

Signature Page for VV-TMF-319540 v1.0